CLINICAL TRIAL: NCT03468595
Title: Clinical Evaluation of Some Local Antimicrobial Agents' Adjunctive Effects On Periodontal Parameters and Halitosis With Subgingival Ultrasonic Instrumentation in Periodontitis Patients: A Randomized Clinical Study
Brief Title: Clinical Evaluation of Some Local Antimicrobial Agents' Adjunctive Effects On Periodontal Parameters and Halitosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Near East University, Turkey (Other)
Responsible Party: Principal Investigator, Hasan Guney YILMAZ, Prof Dr, Near East University, Turkey
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EK-2012-9-51
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Halitosis
Keywords: Listerine, CHX
MeSH Terms: conditions — Halitosis | interventions — Ultrasonography; Emergency Treatment

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- test 1 (Experimental): The treatment of periodontitis was performed with ultrasonic instrumentation (Piezonmaster 700; Electro Medical Systems, Nyon, Switzerland) with CHX (Drogsan, Istanbul, Turkey, 0.2%) was performed at one session for once.
  Interventions: Device: ultrasonic (Piezon Master 700) performed with CHX
- test 2 (Experimental): The treatment of periodontitis was performed with ultrasonic instrumentation (Piezonmaster 700; Electro Medical Systems, Nyon, Switzerland) with Listerine (Johnson & Johnson, Istanbul, Turkey, containing, 21.6% ethanol, 0.092% eucalyptol, 0.064% thymol, 0.042% menthol and 0.06% methyl salicylate) was performed at one session for once.
  Interventions: Device: ultrasonic (Piezon Master 700) performed with Listerine
- control (Active Comparator): The treatment of periodontitis was performed with ultrasonic instrumentation (Piezonmaster 700; Electro Medical Systems, Nyon, Switzerland) with distilled water was performed at one session for once.
  Interventions: Device: ultrasonic (Piezon Master 700) performed with serum

INTERVENTIONS:
Device: ultrasonic (Piezon Master 700) performed with Listerine
  Other Names: EMS, Nyon
  Arms: test 2
Device: ultrasonic (Piezon Master 700) performed with CHX
  Other Names: EMS, Nyon
  Arms: test 1
Device: ultrasonic (Piezon Master 700) performed with serum
  Other Names: EMS, Nyon
  Arms: control

SUMMARY:
The aim of this trial was to establish the clinical efficacy of Listerine and chlorhexidine (CHX) when used as a cooling agent with ultrasonic instrumentation, on periodontal parameters and halitosis.

Ninety patients with periodontal disease participated for the study. Individuals were randomly selected to a control and test groups. At baseline, all subjects completed a questionnaire and carried out an examination. Standard periodontal outcome variables were assessed. For both groups, the plaque index (PI), gingival index (GI), pocket depth (PD), bleeding on probing (BOP) and clinical attachment level (CAL) scores were enrolled at baseline and after 30 days. Volatile sulphur compound (VSC) levels were evaluated by a Halimeter (Interscan Corp., Chatsworth, CA, USA) at baseline (T0), immediately after treatment (T1), and at 7 (T2), 14 (T3) and 30 days (T4).

ELIGIBILITY:
Inclusion Criteria:

* In the present trial, who had periodontitis from patients undergoing periodontal treatment at the Department of Periodontology of our institution

Exclusion Criteria:

* Individuals who presented any systemic disorders which cause halitosis (diabetes mellitus, nephropathy, liver disease, gastrointestinal diseases, respiratory problems), pregnancy or lactation, individuals who had taken antibiotics over the last 6 months or permanently used any drugs, individuals who had any form of periodontal treatment within 6 months prior to the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-03; Primary Completion 2016-09 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Periodontal Pocket Depth (PPD) | 30 day
  PD were evaluated: at the follow-up sessions by the investigator with by marking a point on a 10 mm periodontal probe.

SECONDARY OUTCOMES:
halimeter values | 30 day
  The changes of Volatile Sulphure Compaunds by were evaluated with Halimeter Device at the follow-up sessions by the investigator. The Halimeter reads out in parts-per-billion (ppb) of volatile sulfur compounds.

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Guney YILMAZ, DDS, PhD, Study Director — Near East University, Faculty of Dentistry

IPD SHARING:
Plan to Share IPD: No